CLINICAL TRIAL: NCT03224988
Title: Bilateral Brain Dynamics Supporting Cognition in Normal Aging and Dementia
Brief Title: Bilateral Brain Dynamics in Cognition and Aging
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00085432
Record Dates: First submitted 2017-07-10; First posted 2017-07-21 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease; Aging; MCI
Keywords: Alzheimer's Disease; AD; MCI-AD; MCI; Memory; TMS; Transcranial Magnetic Stimulation; Neuropsychological evaluation; MRI; DTI; EEG
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples were collected on a subset of participants who consented to this additional study component.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Normal Adults
  Interventions: Device: TMS
- MCI Adults
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — A multimodal approach consisting of single pulse TMS, dual-coil TMS, and EEG will be used to examine whether synchronous hemispheric interactions associated with TMS will be present in weighted phase-lag coherence (WPLI), if these measures will be enhanced by in-phase TMS and reduced by counter-phase TMS, and if WPLI will be greater for normal controls than MCI-ADs.

SUMMARY:
This project is focused on the gap in understanding of bilateral brain interactions and their role in helping normative and clinical elderly populations maintain cognitive health. The investigator will focus on investigating this neural mechanism of these interactions and promoting them with a precise application of TMS, in order to test the hypothesis that excitatory interactions between the hemispheres can provide positive outcomes for patients with pre-clinical AD (amnestic Mild Cognitive Impairment or MCI-AD). In Session 1, the investigator will establish the spatial specificity of bilateral brain mechanisms with combination of behavior, TMS, and structural neuroimaging in cortical sites known to be active during memory encoding. In Session 2, the investigator will establish the underlying dynamics of interhemispheric communication using a novel combination of TMS and electroencephalography (EEG) to establish the coordinated activity between the hemispheres; Lastly, in Session 3, the investigator will use the TMS entraining parameters delineated in Aim 2 to promote specific cross-hemispheric communication, applied to participants performing a Picture Encoding task, a general task of memory performance. The outcome of these studies will allow our group to evaluate the strength of this brain stimulation protocol in alleviating age-related and dementia-related cognitive decline, and enable development of novel treatment protocols for dementia in elderly cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent
2. English speaking
3. Signed HIPAA authorization
4. Use of effective method of birth control for women of childbearing capacity

Exclusion Criteria:

1. Current or recent (within the past 6 months) of substance abuse or dependence, excluding nicotine and caffeine (urine test).
2. Current serious medical illness (self report).
3. History of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by TMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator); [TMS Adult Safety Screening (TASS) form].
4. Subjects are unable or unwilling to give informed consent.
5. Diagnosed any Axis I DSM-IV disorder (MINI, DSM-IV)
6. Subjects with a clinically defined neurological disorder including, but not limited to:

   1. Any condition likely to be associated with increased intracranial pressure
   2. Space occupying brain lesion.
   3. History of stroke.
   4. Transient ischemic attack within two years.
   5. Cerebral aneurysm.
   6. Dementia.
   7. Mini Mental Status Exam (MMSE) score of <24.
   8. Parkinson's disease.
   9. Huntington's disease.

   i. Multiple sclerosis.
7. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold.
8. Subjects not willing to tolerate the confinement associated with being in the MRI scanner.
9. Women who are pregnant or breast-feeding (urine test).
10. Blindness.
11. Inability to read or understand English.
12. Intracranial implants, such as:

    1. Cochlear implants;
    2. Aneurysms clips;
    3. Shunts;
    4. Stimulators;
    5. Electrodes;
    6. Cardiac pacemakers;
    7. Vagus Nerve stimulation devices.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Duke Bryan Alzheimer's Disease Research Center Alzheimer's Disease Prevention Registry (ADRC ADPR). Thirty healthy volunteers and thirty MCI-ADs will be recruited.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Establish the structural basis for bilateral brain interactions in healthy older adults. | 2 years
  This will be examined using a Picture Encoding (PE) task in healthy older adults, which will allow identification of spatial brain targets based on the structural pathways connecting left and right DLPFC, ultimately relating the integrity of these pathways based on PE task performance. This Primary Outcome measure will therefore be performance scores (% correct) on this PE task.
Establish the structural basis for bilateral brain interactions in MCI-AD older adults. | 2 years
  This will be examined using a Picture Encoding (PE) task in MCI-AD participants, which will allow identification of spatial brain targets based on the structural pathways connecting left and right DLPFC, ultimately relating the integrity of these pathways based on PE task performance. This Primary Outcome measure will therefore be performance scores (% correct) on this PE task.

SECONDARY OUTCOMES:
Establish the temporal dynamics of cross-hemispheric communication in normal aging using unilateral TMS | 3 years
  An approach consisting of single pulse will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.
Establish the temporal dynamics of cross-hemispheric communication in normal aging using bilateral TMS | 3 years
  An approach consisting of dual-coil TMS will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.
Establish the temporal dynamics of cross-hemispheric communication in normal aging using EEG | 3 years
  An approach consisting of EEG will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.
Establish the temporal dynamics of cross-hemispheric communication in MCI-AD using unilateral TMS | 3 years
  An approach consisting of single pulse will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.
Establish the temporal dynamics of cross-hemispheric communication in MCI-AD using bilateral TMS | 3 years
  An approach consisting of dual-coil TMS will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.
Establish the temporal dynamics of cross-hemispheric communication in MCI-AD using EEG | 3 years
  An approach consisting of EEG will be used to examine synchronous hemispheric interactions associated with TMS. The Secondary Outcome measure will be the weighted phase-lag index (WPLI), which measures the coherence between different brain regions.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Davis, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided